CLINICAL TRIAL: NCT06608472
Title: A Phase III, Randomized, Double-blind, Double-dummy, Active-controlled, Multicenter, Efficacy and Safety Study of a New Fixed-dose Combination of an Angiotensin Receptor Blocker and a Thiazide Diuretic for the Treatment of Essential (primary) Arterial Hypertension
Brief Title: Fixed-dose Combination of an Angiotensin Receptor Blocker and Thiazide Diuretic for Essential Hypertension
Acronym: ATHESA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF187
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Essential Arterial Hypertension
Keywords: hypertension; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N0877 (Experimental): in the test group will be required to take 1 tablet of the test drug N0877. 1 tablet a day for 56 days +/- 4 days.
  Interventions: Drug: N0877
- Benicar HCT® (Active Comparator): in the test group will be required to take 1 tablet of the Benicar HCT®. 1 tablet a day for 56 days +/- 4 days.
  Interventions: Drug: Benicar HCT ® Tablets 40 mg/25 mg

INTERVENTIONS:
Drug: N0877 — 1 tablet of N0877 and 1 tablet of Placebo of Benicar HCT®
  Arms: N0877
Drug: Benicar HCT ® Tablets 40 mg/25 mg — 1 tablet of Benicar HCT® and 1 tablet of Placebo of N0877
  Arms: Benicar HCT®

SUMMARY:
This is a phase III, non-inferiority, randomized, double-blind, double-dummy, active-controlled, multicenter study to compare the efficacy and safety of N0877 versus double combination with already established efficacy on systolic blood pressure (SBP) in the sitting position in the medical office in patients with SAH after 8 weeks of treatment.

DETAILED DESCRIPTION:
This is a phase III, non-inferiority, randomized, double-blind, double-dummy, active-controlled, multicenter study to compare the efficacy and safety of N0877 versus double combination with already established efficacy (olmesartan 40 mg + hydrochlorothiazide 25 mg) in individuals with stage 2 primary arterial hypertension (SBP ≥ 160 ≤ 179 mm Hg or DBP ≥ 100 ≤ 109 mm Hg). This study will be used to support the registration of the new FDC of Eurofarma Laboratórios S.A.

The randomized treatment period aims to demonstrate the non-inferiority of the new combination compared to its comparator on the SBP in patients with SAH in 8 weeks of treatment after randomization.

Throughout the study, the participant must attend to four (04) in-person visits to the research site, being one Screening Visit (VS/V1) throughout the run-in period, one Randomization Visit (VR/V2), one follow-up visit after four (04) weeks (V3), and one Final Visit (VF/V4) after eight (08) weeks of randomized treatment, this being the visit to assess the primary endpoint of the study

ELIGIBILITY:
Inclusion Criteria:

1. Ability to confirm voluntary participation and agree to all purposes of the study, signing and dating the Informed Consent Form in two copies.
2. Age ≥ 18 years.
3. Medical office blood pressure with SBP ≥ 160 mm Hg or DBP ≥ 100 mm Hg without pharmacological treatment or which is not adequately controlled with monotherapy or with a combination of two drugs in which at least one of the drugs is not at the maximum dose.
4. Uncontrolled arterial hypertension (medical office BP with SBP ≥ 140 mm Hg or DBP ≥ 90 mm Hg) after at least two (02) weeks of run-in treatment.
5. Compliance with run-in treatment ≥ 80% and ≤ 120%.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Women in the reproductive age or of childbearing potential who do not agree to use a proven effective contraceptive method, unless they are surgically sterile or expressly declare themselves to be free from the risk of pregnancy because they do not engage in sexual practices or engage in them in a non-reproductive manner.
3. Medical office blood pressure with SBP ≥ 180 mm Hg or DBP ≥ 110 mm mmHg.
4. Resistant hypertension or secondary hypertension of any etiology (including renovascular disease, pheochromocytoma and Cushing's syndrome).
5. Concomitant presence of Coronary Artery Disease, Congestive Heart Failure, Liver Failure and/or Chronic Kidney Disease stage IV or V.
6. History of hypertensive emergencies in the last 6 months.
7. Moderate to severe cardiovascular (acute myocardial infarction or unstable angina, unstable or life-threatening arrhythmia) and/or cerebrovascular events within the last 6 months or any other disorder that in the opinion of the investigator excludes the participant from the study.
8. Participant who is unwilling to switch from hypertension treatment to study medications.
9. 12-lead electrocardiogram (ECG) with any clinically significant abnormality.
10. Drug or alcohol abuse in the last 2 years.
11. Allergic or hypersensitivity reactions to angiotensin II receptor blockers, thiazide diuretics or medication excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2026-11-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in SBP in the sitting position at medical office at week 8 after randomization from baseline | 8 weeks
  To demonstrate the non-inferiority of the N0877 to double combination with an already established profile (olmesartan 40 mg + hydrochlorothiazide 25 mg) on systolic blood pressure (SBP) in the sitting position in the medical office in patients with SAH after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratórios S.A, Itapevi, São Paulo, Brazil